CLINICAL TRIAL: NCT05932849
Title: Benralizumab Patient Access Programme Study: Retrospective, Observational Study in UK Severe Asthma Centres to Describe Patient Characteristics, Treatment Patterns and Outcomes
Brief Title: Benralizumab Patient Access Programme Study: Retrospective Study in UK Severe Asthma Centres
Acronym: BPAP
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00090
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Benralizumab — Patients were initiated on benralizumab as part of routine clinical practice

SUMMARY:
Retrospective secondary data collection observational chart review study. Data collection and analysis will be performed on a cohort of patients who have previously been enrolled on the BPAP. Approximately 300 patients taking part in the BPAP between April 2018 and November 2019 and who meet the eligibility criteria will be recruited to participate in the study.

Data for each participant in the study will be obtained retrospectively with a focus on obtaining data at baseline (12 months prior to first benralizumab dose or at first assessment in the severe asthma center if <12 months), Index date (date of first benralizumab dose) and at least up to 24 months after index date.

Primary Objectives

* To describe baseline demographic and clinical characteristics of severe eosinophilic asthma patients enrolled in the BPAP
* To describe background treatment patterns of severe eosinophilic asthma patients at baseline and after benralizumab initiation

Secondary Objectives:

* To describe clinical outcomes after initiation of benralizumab therapy in severe eosinophilic asthma patients treated with benralizumab at 12 and 24 months
* To describe patients' adherence to benralizumab, persistence and discontinuation rates and reasons for discontinuation at 12 and 24 months

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled on the BPAP between April 2018 and November 2019
* Patients who have at least 1 benralizumab injection and with at least 3 months followup data from the time of enrolment into the BPAP
* Patients initiated on benralizumab outside of the BPAP by October 30, 2019.
* Where CRO employees conduct the data extraction, patients must be able and willing to give informed consent to participate in the study

Exclusion Criteria:

* Currently receiving benralizumab or any other biologic drug for the treatment of asthma in a clinical trial
* Refusal or inability to provide informed consent where the CRO will be collecting the data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe eosinophilic asthma patients enrolled in the benralizumab patient access programme in UK severe centres. Patients will have had their first benralizumab dose between April 2018 and November 2019 and data will be collected retrospectively between May 2019 and October 2021.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Baseline annual exacerbation rate | -12 to 0 months
  Baseline frequency and annualized rate of asthma exacerbations by severity levels
Maintenance OCS dose during baseline | -12 to 0 months
  Maintenance OCS: frequency of patients on mOCS, dosage (for patients on mOCS), annualized cumulative dose

SECONDARY OUTCOMES:
Annualised exacerbation rate (AER) | 12 months
  AER at 12 months
Annualised exacerbation rate (AER) | 24 months
  AER at 24 months
FEV1 | 12 months
  change in lung function from baseline
FEV1 | 24 months
  change in lung function from baseline
ACQ-6 | 12 months
  Change in asthma control (ACQ-6) score from baseline
ACQ-6 | 24 months
  Change in asthma control (ACQ-6) score from baseline
AQLQ(S)+12 | 12 months
  Change in asthma quality of life (AQLQ) from baseline
AQLQ(S)+12 | 24 months
  Change in asthma quality of life (AQLQ) from baseline
Eosinophil count | 12 months
  Mean change in eosinophil count from baseline
Eosinophil count | 24 months
  Mean change in eosinophil count from baseline
mOCS dose | 12 months
  Percentage change in daily OCS dose, Percentage of patients with OCS <=5mg/day (only for those patients that at baseline had a daily dose >5mg/d)
mOCS dose | 24 months
  Percentage change in daily OCS dose, Percentage of patients with OCS <=5mg/day (only for those patients that at baseline had a daily dose >5mg/d)
Treatment persistence | 24 months
  Proportion of patients discontinuing benralizumab and proportion by reason for discontinuation
Adherence to scheduled injections | 24 months
  * Frequency of patients taking infections on schedule
  * Frequency of patients taking injection within +/- 3 days injection window in an observation period
  * Time between injections

CONTACTS AND LOCATIONS:
Overall Officials: David J Jackson, MRCP MSc PhD, Principal Investigator — Guy's & St Thomas' NHS Trust
Locations (8):
- United Kingdom (8):
  - Addenbrookes Hospital, Cambridge
  - Castle Hill Hospital, Hull
  - St James's University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Guy's Hospital, London
  - Royal Brompton Hospital, London
  - St Bartholomew's Hospital, London
  - Southampton General Hospital, Southampton

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00090&attachmentIdentifier=98d5d97e-ba89-4244-8551-245aa79edf0a&fileName=BPAPII_AZ_CSR_Synopsis_V1.0_06Nov2023_Redacted.pdf&versionIdentifier=